CLINICAL TRIAL: NCT00553020
Title: Assessment of Duration of Metabolic Effect of a Single Bolus of Subcutaneous Injected Lantus Compared to NPH-Insulin(Protaphan)in Patients With Type 2 Diabetes
Brief Title: Assessment of Duration of Metabolic Effect of a Single Bolus of sc Injected Lantus Compared to NPH Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HOE901_4050
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: Insulin glargine — Lantus (commercial formulation, Reference):
  10 mL vials (100 IU/mL) solution Dose: 0.3 IU per kg BW injected subcutaneously in the patients usual injection site (either abdomen or thigh)
  NPH-insulin (Protaphan) (Test):
  10 mL vials (100 IU/mL) solution Dose: 0.3 IU per kg BW injected subcutaneously in the patients usual injection site (either abdomen or thigh)

SUMMARY:
To assess the duration of the metabolic effect of a sc injected single dose of either insulin glargine (LantusT) or NPH-insulin (ProtaphanT) on blood glucose control in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus of either gender as defined by the American Diabetes Association (3) for more than 6 months
* BMI (as defined in Appendix A of the protocol) between 28 kg/mý and 32 kg/mý (before implementation of Amendment 1) or between 26 kg/mý and 34 kg/mý (after implementation of Amendment 1)
* Having required treatment with insulin for at least 6 months
* Stable glycemic control with glycohemoglobin (HbA1c) >7.5% and <9.5% (before implementation of Amendment 1) or >7.0% and <9.5% (after implementation of Amendment 1
* Fasting serum C-peptide >0.2 pmol/mL. According to Amendment 3, five additional subjects with "low" (defined as less than or equal to 0.4 pmol/mL) and 5 subjects with "high" (defined as >0.4 pmol/mL) fasting C-peptide were to be enrolled.
* Negative pregnancy test in female subjects of childbearing potential (only for those who were not surgically sterile or who were less than 2 years postmenopausal) at the beginning of the study
* No findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and muscular-skeletal system) which were clinically relevant and interfering with the conduct of the study
* Normal ECG, blood pressure, pulse rate and core body temperature unless the investigator considered an abnormality to be clinically irrelevant and not interfering with the conduct of the study

Exclusion Criteria:

* Subjects with "brittle" diabetes or predisposition to severe hypoglycemia, e.g. 2 or more severe hypoglycemic episodes (i.e. requiring assistance of another person) within the past year, or any hospitalization or emergency room visit due to poor diabetic control within the past 6 months
* Subjects who had been treated with insulin with a total insulin dose of >1.5 IU/kg/day
* Pregnant and nursing women
* Female subjects of childbearing potential (those who are not surgically sterile or who are less than 2 years postmenopausal) unwilling or unable to use reliable contraceptive measures. Reliable contraceptive measures included the following: systemic contraceptive (oral, implant, injection), diaphragm with intravaginal spermicide, cervical cap, intrauterine device, or condom with spermicide.
* Any condition requiring the regular use of any medication if the regular use of this medication interfered with the study conduct
* Abuse of alcoholic beverages (as defined in Appendix B of the protocol)
* Treatment with oral antidiabetic drugs within the last 4 weeks
* Treatment in the previous 3 months with any drug known to have a well-defined potential for toxicity concerning vital organs
* Symptoms of any major internal medical disease in the 4 weeks before the study which, according to the investigator's opinion, could interfere with the purposes of the study
* History of hypersensitivity to any drugs that have a similar chemical structure to the study drug
* History or presence of gastrointestinal, liver, or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Blood donation during the previous 3 months
* Positive HIV- or hepatitis B/C-test
* Progressive fatal disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-04; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To assess the duration of the metabolic effect of a sc injected single dose of either insulin glargine (LantusT) or NPH-insulin (ProtaphanT) on blood glucose control in patients with type 2 diabetes | during the study conduct

SECONDARY OUTCOMES:
To evaluate the effect of insulin glargine (LantusT) and NPH-insulin (ProtaphanT) on suppression of endogenous glucose production, endogenous insulin secretion, and lipolysis | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Karim El-Haschimi, Study Director — Sanofi